CLINICAL TRIAL: NCT05062421
Title: Persistence of Biological Treatment and Inhibitors of Jak Kinases in Habitual Clinical Practice in Patients With Rheumatoid Arthritis. Influence of the Comorbidities.
Brief Title: Persistence of Biological Treatment and Inhibitors of Jak Kinases in Patients With Rheumatoid Arthritis.
Acronym: Arthritis
Status: Recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-FME-2020-01
Record Dates: First submitted 2021-09-10; First posted 2021-09-30 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-04

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cases 1: Patients treated with JAK-type kinase inhibitors.
- Cases 2: Patients treated with monoclonal antibodies against TNF.
- Cases 3: Patients treated with soluble receptor against TNF.
- Cases 4: Patients treated with FAME group biosimilars.
- Cases 5: Patients treated with rituximab.
- Cases 6: Patients treated with abatacept.
- Cases 7: Patients treated with drugs that block the IL6.

SUMMARY:
One-center observational study aimed at determining the survival of patients with rheumatoid arthritis treated with targeted synthetic disease-modifying drugs (FAMEsd) and biologic disease-modifying drugs (FAMEb).

These patients will be administered a series of medications and a follow-up will be carried out to analyze their evolution.

DETAILED DESCRIPTION:
One-center observational study aimed at determining the survival of patients with rheumatoid arthritis treated with targeted synthetic disease-modifying drugs (FAMEsd) and biologic disease-modifying drugs (FAMEb).

The drugs to be administered to patients are:

* JAK-type kinase inhibitors.
* Monoclonal antibodies against TNF.
* Soluble receptor against TNF.
* Biosimilar FAMEb.
* Rituximab.
* Abatacept.
* Drugs that block IL6.

A follow-up will be carried out at 12, 24, 48, 60, 72 and 84 months from the start of treatment, to analyze how the patient's health improves.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* With a diagnosis of Adult Rheumatoid Arthritis according to the 2010 ACR / EULAR criteria.
* Who have received at least one of the doses of the study drugs.
* In follow-up in the consultations of the UGC of Rheumatology of the HUVM.
* With at least two complete evaluations (baseline and final) of clinical variables.

Exclusion Criteria:

* Patients where the medical records lack sufficient baseline and final variables to perform the analysis.
* Patients in whom more than 50% of the variables to be collected are missing in the data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 years diagnosed with rheumatoid arthritis, who have been under treatment with at least one dose of the study drugs, whose treatment is followed by the rheumatology unit.
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival study | Up to 60 weeks
  To know the survival at 12, 24, 48, 60, 72 and 84 months to the synthetic directed anti-rheumatic drugs, disease modifiers (FAMEsd) and the biological disease modifying anti-rheumatic drugs (FAMEb) in patients with rheumatoid arthritis treated in routine.

SECONDARY OUTCOMES:
Study of clinical characteristics. | Up to 60 weeks
  To know the sociodemographic and clinical characteristics of the patients who receive FAMEsd and FAMEb in routine clinical practice at the HUVM.
Measure of the influence of comorbidities. | Up to 60 weeks
  To assess the influence of comorbidities on drug persistence.
Number of participants who discontinued treatment due to serious adverse effects. | Up to 60 weeks
  Failure due to serious adverse events, adverse events of special interest, emerging adverse events and minor adverse events that require discontinuation of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Estela Hernández Cruz, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen macarena, Seville, Spain